CLINICAL TRIAL: NCT04130854
Title: INNATE: Immunotherapy During Neoadjuvant Therapy for Rectal Cancer, a Phase II Randomized Multi-center Trial With and Without APX005M, an Anti-CD40 Agonist
Brief Title: INNATE: Immunotherapy During Neoadjuvant Therapy for Rectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Apexigen America, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Todd Aguilera, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2019-1492; 5R01CA283953-03 (NIH)
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Rectal Adenocarcinoma
MeSH Terms: interventions — sotigalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- APX005M on day 3 of RT & day 3 of cycles 1-5 of mFOLFOX (Experimental): On Day 3 of Cycles 1-5 of each mFOLFOX treatment, participants will receive another dose of APX005M. The sequence of administration of APX005M in combination with mFOLFOX. In Cycle 6, participants will receive only mFOLFOX. After completing the last planned dose of mFOLFOX, participants will be considered off-protocol directed therapy and undergo planned TME, per institutional standards, and proceed to the follow-up portion of this study.
  Interventions: Drug: APX005M, mFOLFOX, and Radiation Therapy 5Gy x 5 days
- Radiation Therapy 5Gy x 5 days, mFOLFOX (Active Comparator): Participants randomized to Arm 2 will receive short-course RT and mFOLFOX regimen, except that participants will not receive any of the study drug. After completing the last planned dose of mFOLFOX, participants will be considered off-protocol directed therapy and undergo planned TME, per institutional standards, and proceed to the follow-up portion of this study.
  Interventions: Drug: mFOLFOX and Radiation Therapy 5Gy x 5 days

INTERVENTIONS:
Drug: APX005M, mFOLFOX, and Radiation Therapy 5Gy x 5 days — 1. APX005M 0.3mg/kg intravenously on day 3 of radiation and on day 3 of cycles 1-5 of mFOLFOX
  2. Short course radiation therapy 5 Gy x 5 days
  3. Oxaliplatin 85mg/m2 intravenous day 1 of each cycle
  4. Leucovorin 400mg/m2 IV Day 1 of each cycle
  5. 5-FU 2400 mg/m2 continuous infusion over 46 hours of each cycle
  Arms: APX005M on day 3 of RT & day 3 of cycles 1-5 of mFOLFOX
Drug: mFOLFOX and Radiation Therapy 5Gy x 5 days — 1. Short course radiation therapy 5 Gy x 5 days
  2. Oxaliplatin 85mg/m2 intravenous day 1 of each cycle
  3. Leucovorin 400mg/m2 IV Day 1 of each cycle
  4. 5-FU 2400 mg/m2 continuous infusion over 46 hours of each cycle
  Arms: Radiation Therapy 5Gy x 5 days, mFOLFOX

SUMMARY:
Determine the complete pathologic complete response (pCR) rate in patients with locally advanced rectal adenocarcinoma.

DETAILED DESCRIPTION:
A phase II randomized trial 3:2 with short course radiotherapy followed by mFOLFOX chemotherapy prior to trans abdominal resection with or without an antiCD40 agonist antibody (APX005M). There will be continuous safety assessment for at least 6 patients. Planned accrual of 58 patients. An interim analysis after 30 patients have completed treatment and there will be early stopping criteria for futility or efficacy. Short course radiotherapy will consist of 5Gy x 5 to the pelvis and patients on APX005M arm will receive one infusion during radiotherapy course, have a two week break, then start FOLFOX with APX005M in conjunction with five out of six cycles of chemotherapy. Patients will be restaged and then undergo definitive surgery.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age. Both men and women and members of all races and ethnic groups will be included.
2. Willing and able to provide written informed consent
3. Pathologic diagnosis of rectal adenocarcinoma
4. Stage III or Stage II with at least 1 of the following high-risk features:

   * Distal (<1cm from anal ring)
   * cT4 or within 3mm of MR fascia
   * Not candidate for sphincter preservation
   * Extramural venous invasion
5. No prior treatment for rectal adenocarcinoma
6. Eastern Cooperative Group (ECOG) performance status of 0-1.
7. Laboratory values supporting acceptable organ and marrow function within 21 days of eligibility confirmation. Defined as follows:

   * WBC ≥ 3,000/mL;
   * ANC WBC ≥ 1,500/mL;
   * PLT ≥ 100,000/mL;
   * T Bili ≤ 1.5 x upper limit of normal (ULN);
   * AST/ALT ≤ 2.5 x ULN;
   * Creatinine ≤ 1.5 times upper limit of normal or calculated creatinine clearance > 45 mL/min per Cockcroft-Gault equation.
8. Female participants of childbearing potential (FOCBP) must have a negative serum or urine pregnancy test (per institutional standards) within 72 hours prior to the start of study drug.

   FOCBP must agree to use highly-effective method(s) of contraception (Appendix A) during the study and for 90 days after the last dose of study drugs.

   FOCBP are those who have not been surgically sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy) or have not been free from menses for >1 year without an alternative medical cause.
9. Male participants must agree to use an adequate method of contraception (Appendix A) starting with the first dose of study therapy through 90 days after the last dose of study drugs.

Exclusion Criteria:

1. Distant nodal disease (retroperitoneal nodes) including inguinal nodes, or any metastatic disease by CT or PET
2. Prior RT to the pelvis.
3. Uncontrolled comorbid illness or condition including an active infection, congestive heart failure, unstable angina, cardiac arrhythmia, or psychiatric illness that would limit compliance with the study requirements.
4. Prior treatment with any anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
5. Any positive history for HIV/AIDS, HTLV, hepatitis B or hepatitis C virus indicating acute or chronic infection.
6. Any active known or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
7. Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to the first dose of study drug. Inhaled steroids and adrenal replacement steroid doses up to 10 mg daily prednisone equivalent are permitted (although not encouraged) in the absence of active autoimmune disease.
8. Malignancy in the past 3 years that required active treatment except locally curable cancers or cancers deemed by the treating physicians to not impact the subject's survival duration.
9. Participants receiving any other investigational agent, standard antineoplastic agents, or immunosuppressive agents.
10. Known history of interstitial lung disease.
11. Received live vaccine within 6 weeks prior to randomization.
12. Psychiatric illness/social situations that would limit consenting and compliance with study requirements.
13. Participants who are pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
14. Patient is not a candidate for the full treatment regimen.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2020-04-24 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response Rate | At time of surgery
  The primary objective of this study is to determine the pathologic complete response (pCR) rate of the combined treatment modality.

SECONDARY OUTCOMES:
Overall Survival | 3 years
  To evaluate overall survival (OS), defined as the time between date of randomization and the date of death due to any cause.
Toxicity analysis | 3 years
  To evaluate toxicity analysis comparing the experimental from the standard arm measured according to CTCAE v5.0.
Disease free survival | 3 years
  To evaluate the disease free survival (DFS) and patterns of failure at three years. DFS is defined as the time between the date of definitive surgery and the first date of documented disease progression or death.

OTHER OUTCOMES:
Exploratory Immunological Response | 3 years
  To evaluate the immunologic response surrogates for patients tissue is obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Aguilera, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (4):
- United States (4):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Wake Forest Baptist Health Sciences, Winston-Salem, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Undecided